CLINICAL TRIAL: NCT05859230
Title: A Study of a Probiotic (Lacticaseibacillus Paracasei Strain Shirota) Intervention on Gut Microbiota and Cognitive Functioning in Older Adults With Mild Cognitive Impairment
Brief Title: Probiotic Intervention on Gut Microbiota and Cognitive Functioning in Older Adults With a Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Rathi Mahendran, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-696
Record Dates: First submitted 2023-01-04; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Probiotic; Gut microbiota; Mild cognitive impairment; Older adults; Intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The probiotic drink study group (Experimental): Older adults between 60-90 years of age, diagnosed with Mild Cognitive Impairment, will participate in an 18-week long study consisting of the probiotic drink consumption for 12 weeks, followed by a 6-week follow-up period.
  Interventions: Dietary Supplement: Experimental: The probiotic drink study group
- The placebo drink study group (Placebo Comparator): The older adults between 60-90 years of age, diagnosed Mild Cognitive Impairment, participate in the total 18-week longed study consisting of the placebo milk drink consumption for 12 weeks, followed by a 6-week follow-up period.
  Interventions: Dietary Supplement: Placebo Comparator: The placebo drink study group

INTERVENTIONS:
Dietary Supplement: Experimental: The probiotic drink study group — The 100 ml volume of milk drink containing 10 billion Lacticaseibacillus paracasei strain Shirota is consumed once a day for 12-week intervention period, followed by a 6-week follow-up period. The intervention is double-blinded by study team members and subjects. The milk drink bottles are coded by the manufacturing company.
  Arms: The probiotic drink study group
Dietary Supplement: Placebo Comparator: The placebo drink study group — The 100 ml volume of milk drink without containing Lacticaseibacillus paracasei strain Shirota is consumed once a day for 12-week intervention period, followed by a 6-week follow-up period. The intervention is double-blinded to study team members and subjects. The milk drink bottles are coded by the manufacturing company.
  Arms: The placebo drink study group

SUMMARY:
Recent studies suggest that gut microbiota is linked to cognitive performance and modulating gut microbiota is a safe and promising approach to enhance cognition. The limited studies in the area of probiotics for cognitive impairment in early stages warrant further research. In this feasibility study, we will examine the effects of probiotic consumption in older adults with mild cognitive impairment (MCI), on gut microbiota and cognition via microbiota composition, inflammatory, immune, and bacterial metabolite mechanisms, using neuropsychological tests. The single probiotic contains the Lacticaseibacillus paracasei strain Shirota (LcS), with proven efficacy in various health conditions as well as in stress, sleep, and mood disorders; but to our knowledge, it has not been rigorously examined in early stages of cognitive impairment. After 12 weeks of the randomized, double-blinded probiotic/placebo intervention, we hypothesize that the changes in the composition of gut microbiota, short-chain fatty acids, and the inflammatory/immunological markers, could improve functional connectivity and cognition.

DETAILED DESCRIPTION:
The 18-week study consists of a 12-week intervention period and a 6-week follow-up period. Chinese older adults between 60 and 90 years of age and known to have Mild Cognitive Impairment and agree to participate in this study will be screened for eligibility and then randomized into 2 arms. Subjects will be recruited from current ongoing studies from NUS under NUS-IRB registration and the study posters at the National University Hospital clinic. Those participants who consented to be contacted by the study team to participate in further research activities and with a diagnosis of Mild Cognitive Impairment will be first contacted by research team members from that study. All of them will be briefly informed about this intervention study and asked if they agree to be contacted for more information. Written informed consent will be taken for the intervention groups. Subject screening and enrolment will be documented by the study team using a screening log. Drop-out and screen failures will be documented.

The probiotic and placebo drink bottles will be coded by the manufacturing company and delivered with a sealed envelope containing the code. Subjects who meet the study eligibility criteria will be randomly assigned using online study randomization software to one of the coded groups corresponding to the probiotic or placebo study groups. Both Study team members and subjects will be blinded to the intervention. The study product codes/blinding will be broken either: (1) at the end of the study for analysis, or (2) in the event of a serious adverse event as deemed necessary by the study team.

Subjects should drink the study product (active interventional probiotic or placebo depending on randomization) 1 bottle per day at breakfast for 12 weeks. Subjects will be given the study product at 2 weekly intervals till the study ends. Subjects who have successfully completed the product consumption period will enter the follow-up period, during which they will continue their normal diet with the exception of fermented dairy products (such as yogurt, Lactobacillus beverages and probiotic supplements). The safety and tolerability parameter will be reports of any adverse events related to the study intervention between the start at Week 0 till the end of the study at Week 18. These will include reports of mild events such as any discomforts (vomiting, bloated sensation, changes in defecation frequency, etc.). Compliance based on the study product consumed and intake of other dairy-fermented milk will be performed at each scheduled visit for all subjects. The study team will review the subject diaries together with the subjects in order to check compliance. Subjects will also be asked to bring empty bottles every 2 weeks when they come to collect another 2 weeks of the intervention product. Compliance will be reinforced at each study visit.

The primary parameter is the change in gut microbiota composition from before to after 12 weeks of probiotic consumption and after stopping probiotic use for 6 weeks (at Week 0, 6, 12 and 18 of the study period). The secondary study parameters will be the changes in cognition at 0, 12 and 18 weeks of the study period, and immune and inflammatory blood markers, and cortisol levels and changes in fecal short-chain fatty acid levels at 0, 6, 12 and 18 of the study period. Basic demographic data, medical history, medications and consumption of diets will be assessed before probiotic consumption.

The fecal sample collection by a subject will be in special containers at home. Two tubes will be required at each time point. The sampling kit will be provided by the study team. Instructions for fecal sample collection will be provided to the subjects by the study team on Visit 1 (screening) for the subsequent visits. Individual samples will be weighed and recorded. The fecal DNA extraction and 16s rRNA sequencing will proceed with the fecal samples from the OMNIgene GUT tube. The analysis will be performed by the NovaSeq 16srRNA amplicon sequencing method. Fecal SCFAs analysis will be performed by Gas chromatography-triple quadrupole mass spectrometer with the fecal samples from OMNI-MET tube.

Two tubes of blood will be collected from each subject at each time point: One tube with 3ml of blood for serum cortisol estimation, and 3mls of blood for the whole blood immune activation assays and for circulating inflammatory marker analysis. Fasting blood is required for cortisol estimation and so blood collection will be scheduled between 9:00 and 11:00 a.m. to minimize diurnal variation in cortisol. The serum cortisol level will be tested by the Electrochemiluminescence immunoassay. The whole blood samples will be centrifuged at 1650 × g for 25 min at room temperature to obtain plasma. The plasma samples will then be stored in aliquots at -80° C until further analyses. The whole blood will be stimulated by Toll-like receptors TLR2 and TLR4 agonists for 48 hours. The supernatant will be collected and aliquot and stored at -80°C. After sample collections from all the time points are completed, all samples for the same participants from different time points will be measured on the same day and on the same plates, to avoid batch effects. The cytokines analyzed will be IL-1β, IL-6, IL-10, IL-8 and TNF- alpha using commercially available enzyme-linked immunosorbent assay (ELISA) kits. All the experiments will be performed as per the instructions of the respective manufacturers of the kits. The stored plasma will be analyzed for 45 biomarkers (cytokines and chemokines) using the Proximity Extension Assay.

This neurocognitive battery of tests has been utilized and validated in the Singaporean population. The tests evaluate various cognitive functions, including attention, learning, memory, speed, and executive function. The tests included Rey Auditory Verbal Learning Test (RAVLT), Digit Span task, Color trails tests, Blcok design and Semantic Verbal fluency test, and Stroop test.

Data collected from demographics, questionnaires, Neuropsychological tests and collected samples will be summarized using descriptive techniques. Summary statistics (mean, standard deviation) will be presented for continuous variables (and their changes from baseline and absolute values at each time point). Counts and percentages will be presented for categorical variables. Where appropriate, the presentation of results will include plot and confidence intervals. Multivariate data analyses of cognitive and biomarker outcomes will be performed using SPSS and R.

ELIGIBILITY:
Inclusion Criteria:

1. able to commit to the 18-week study;
2. aged between 60 and 90 years;
3. has Mild Cognitive Impairment; (Individuals with MCI have the mental capacity to provide their informed consent to participate in research);
4. no regular consumption of fermented dairy products (such as yogurt, Lactobacillus beverages, and probiotic supplements); other fermented products such as cheese, kimchi, miso, soy sauce, and fish sauce can be consumed in small amounts (for example as additives in cooking). If subjects are consuming fermented dairy products regularly and are willing to stop, they can be enrolled after 2 weeks;
5. willing to consume the study product (probiotic /placebo) for 12 weeks and provide the blood and fecal samples of four time points;
6. no history of Diabetes and no history of Head Injury, Seizures or Stroke and are able to travel independently to the study site;
7. other medical co-morbidity, if present, is stable, with no history of change of medications in the last 2 weeks; not taking antibiotics or gastrointestinal medications in the last 2 weeks;
8. no known psychiatric illnesses and not receiving psychotropic medication;
9. bowel movement not less than three times a week;
10. has not participated in any other interventional research in the last 3 months;
11. are not lactose intolerant and have no milk allergy.

Exclusion Criteria:

1. unable to commit to the 18-week study;
2. age below 60 years or above 90 years;
3. does not have Mild Cognitive Impairment or has Dementia;
4. those with a history of Diabetes or history of Head Injury, Seizures and Stroke, and those who for any physical reason cannot come to the study site for assessments;
5. presence of other unstable medical co-morbidity, history of recent change of medications in the last 2 weeks or taking antibiotics or gastrointestinal medications in the 2 weeks prior to the study;
6. those with a psychiatric illness (e.g., Depression or Anxiety) and are receiving psychotropic medication;
7. participation in any interventional research in the last 3 months;
8. regular consumption of fermented dairy products (such as yogurt, Lactobacillus beverages, and probiotic supplements) and other fermented products (such as cheese, kimchi, miso, soy sauce, and fish sauce) in large amounts and are not willing to stop these for 2 weeks before enrolment;
9. not willing to consume the study product (probiotic/placebo) for 12 weeks and provide the blood and fecal samples at four time points;
10. those with bowel movement less than three times a week;
11. have a history of lactose intolerance and/or milk allergies.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in composition of gut microbiota after probiotic and placebo intervention | Baseline, 6 weeks, 12 weeks of intervention and 6 weeks follow-up
  Changes in gut microbiota composition in their abundances using 16s rRNA DNA sequencing method before the intervention, at 6 weeks and 12 weeks after the intervention and at 6 weeks follow-up will be analyzed.

SECONDARY OUTCOMES:
Changes in verbal learning and memory function of neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in learning and memory function of the neurocognitive tests before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes Rey's auditory verbal learning test (RAVLT) which measures immediate and delayed memory and recognition memory. The individual raw numbers of correctly recalled and recognized (0-15) will be analyzed and compared.
Changes in attention and verbal working memory function of neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in attention and verbal working memory function of neurocognitive tests before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes the Digit Span task. The individual raw numbers of scores (0-16) will be analyzed and compared.
Changes in sustained attention and reasoning function by color trails neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in attention and reasoning function of neurocognitive tests before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes the Color Trails test. The individual time taken in seconds will be analyzed and compared.
Changes in sustained attention and reasoning function by Stroop test of neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in attention and reasoning function of neurocognitive tests before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes the Stroop test. The individual time taken in seconds will be analyzed and compared.
Changes in language, lexical knowledge and semantic memory function of neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in language and semantic memory function of neurocognitive tests before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes semantic verbal fluency (animals) tests. The individual raw numbers of animals correctly named (0-40) will be analyzed and compared.
Changes in visuospatial, organizational non-verbal processing function of neurocognitive assessment after probiotic and placebo intervention | Baseline, 12 weeks of intervention and 6 weeks follow-up
  Changes in visuospatial, organizational non-verbal processing function of the neurocognitive test before the intervention, at 12 weeks after the intervention, and at 6 weeks follow-up will be analyzed. The assessment of the function includes total Block design scores. The individual raw numbers of scores (eg. 0-68) will be analyzed and compared.
Changes in plasma immune and inflammatory markers after probiotic and placebo intervention | Baseline, 6 weeks, 12 weeks of intervention and 6 weeks follow-up
  The plasma immune and inflammatory markers such as 45 plasma cytokines/chemokines levels (pg/ml) panel will be measured using the proximity extension assay (PEA) before the intervention, at 6 and 12 weeks after the intervention, and at 6 weeks follow-up.
Changes in blood immune and inflammatory markers in-vitro stimulation by toll-like receptors agonists after probiotic and placebo intervention | Baseline, 6 weeks, 12 weeks of intervention and 6 weeks follow-up
  Whole blood will be stimulated with toll-like receptors 2 and 4 agonists after the collection of blood. The cytokines IL-1 beta, IL-6, IL-10, IL-8 and TNF-alpha will be analyzed using the Enzyme-linked immunosorbent assay (ELISA) method and reported their levels in pg/ml.
Changes in blood cortisol levels after probiotic and placebo intervention | Baseline, 6 weeks, 12 weeks of intervention and 6 weeks follow-up
  The blood cortisol levels (nmol/L) will be measured using an Electrochemiluminescence immunoassay before the intervention, at 6 and 12 weeks after the intervention, and at 6 weeks follow-up.
Changes in fecal short-chain fatty acids after probiotic and placebo intervention | Baseline, 6 weeks, 12 weeks of intervention and 6 weeks follow-up
  The fecal short-chain fatty acids (uM/g of feces) will be measured using a Gas chromatography-triple quadrupole mass spectrometer (GC-MS) in fecal supernatants at baseline, at 6 and 12 weeks after the intervention, and at 6 weeks follow-up.

OTHER OUTCOMES:
Differences in frequency of consumption of diets between probiotic and placebo intervention groups at baseline | Baseline
  Dietary questionnaires will be recorded at baseline before the intervention. The frequency of consumption of diets per day in terms of carbohydrates, proteins, vegetables, fruits, fermented foods and dairy, nuts, fast foods, beverages, desserts, and local snacks will be analyzed in two intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, M.B.,B.S, Principal Investigator — National University of Singapore; Su Hui Ho, M.B.,B.S, Principal Investigator — National University of Singapore
Locations (1):
- Hannah Active Ageing Centre, Singapore, Singapore

REFERENCES:
- [Background] Khine WWT, Voong ML, Ng TKS, Feng L, Rane GA, Kumar AP, Kua EH, Mahendran R, Mahendran R, Lee YK. Mental awareness improved mild cognitive impairment and modulated gut microbiome. Aging (Albany NY). 2020 Dec 9;12(23):24371-24393. doi: 10.18632/aging.202277. Epub 2020 Dec 9. PMID 33318317
- [Background] Hori T, Matsuda K, Oishi K. Probiotics: A Dietary Factor to Modulate the Gut Microbiome, Host Immune System, and Gut-Brain Interaction. Microorganisms. 2020 Sep 11;8(9):1401. doi: 10.3390/microorganisms8091401. PMID 32933067
- [Result] Kailasapathy K, Chin J. Survival and therapeutic potential of probiotic organisms with reference to Lactobacillus acidophilus and Bifidobacterium spp. Immunol Cell Biol. 2000 Feb;78(1):80-8. doi: 10.1046/j.1440-1711.2000.00886.x. PMID 10651933